CLINICAL TRIAL: NCT07072234
Title: Phase I Study of Allogeneic Transforming Growth Factor-beta Receptor Type 2 Knockout CD70 CAR NK Cells in Treatment Refractory Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0508; NCI-2025-04901 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Clear Cell Carcinoma; Phase 1; Growth Factor
MeSH Terms: conditions — Adenocarcinoma, Clear Cell | interventions — Dexamethasone; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose-optimization phase (Experimental)
  Interventions: Drug: Lymphodepleting chemotherapy; Drug: Dexamethasone; Drug: Fludarabine; Drug: Cyclophosphamate; Drug: TGFBR-2 KO CD70 CAR NK
- Dose-expansion phase (Experimental)
  Interventions: Drug: Lymphodepleting chemotherapy; Drug: Dexamethasone; Drug: Fludarabine; Drug: Cyclophosphamate; Drug: TGFBR-2 KO CD70 CAR NK

INTERVENTIONS:
Drug: Lymphodepleting chemotherapy — Given by IV
Drug: Dexamethasone — Given PO
Drug: Fludarabine — Given by IV
Drug: Cyclophosphamate — Given by IV
Drug: TGFBR-2 KO CD70 CAR NK — Given by IV

SUMMARY:
Testing an investigational cancer therapy called TGFBR-2 KO CD70 CAR NK cell therapy.

DETAILED DESCRIPTION:
Primary Objective • To determine the safety, tolerability, maximum tolerated dose (MTD), and optimal celldose (OCD) of chimeric antigen receptor TGFBR-2 KO CD70 CAR NK cells in participants with advanced ccRCC.

Secondary Objectives

• To determine the antitumor activity of TGFBR-2 KO CD70 CAR NK cells. Although the clinical benefit of TGFBR-2 KO CD70 CAR NK cells has not yet been established in ccRCC, the intent of offering this treatment is to provide a possible therapeutic benefit and thus, the participants will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability.

ELIGIBILITY:
Eligibility Criteria

* Participants must have histologically confirmed ccRCC that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Confirmation of CD70 expression ≥ 10% by immunohistochemistry staining of the participants primary renal tumor or a metastatic lesion biopsy specimen will be required for enrollment in the study.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
* Participants must have previously received treatment with at least one ICI and one TKI. Participants must have had unequivocal disease progression on ICI treatment.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of CD70 TGFβR-2 knockout CAR NK cells in Participants <18 years of age, children are excluded from this study.
* Participants must be at least 2 weeks from last cytotoxic chemotherapy, tyrosine kinas inhibitors or other targeted therapies at the time of administration of lymphodepleting chemotherapy.
* Participants must be at least 3 months from any cell therapy for malignancy.
* Localized radiotherapy to 1 or more disease sites is allowed prior to the lymphodepleting chemotherapy, provided that there are additional measurable non-irradiated disease sites.
* Eastern Cooperative Oncology Group performance status 0 or 1 (Performance level as measured by Karnofsky for Participants > 16 years of age.
* Adequate organ function at screening, as defined by the following:

  * Renal: Serum creatinine ≤ 1.5 mg/dL or estimated glomerular filtration rate (Chronic Kidney Disease Epidemiology Collaboration equation) ≥30 ml/min/1.73 m2o Hepatic: alanine transaminase (ALT)/aspartate transaminase (AST) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5 x ULN if documented liver metastases, total bilirubin ≤ 1.5 mg/dL or ≤ 3.0 mg/dL for Participants with Gilbert's Syndrome. No history of liver cirrhosis.
  * Cardiac: Cardiac ejection fraction ≥ 40%, no clinically significant pericardial effusion as determined by echocardiogram (ECHO) or multigated acquisition (MUGA) scan, and no symptomatic cardiac disease or history of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
  * Pulmonary: No clinically significant pleural effusion (per principal investigator [PI] judgement), and baseline oxygen saturation ≥ 92% on room air. Subjects with active interstitial lung disease (ILD)/pneumonitis requiring treatment with systemic steroids will be excluded.
* Hematological: absolute neutrophil count (ANC) ≥ 1000/mm3, platelet count ≥ 75,000/mm3, and hemoglobin ≥ 8 g/dL.

  o Coagulation: International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 ULN. Participants on therapeutic doses of anticoagulation medication must have INR and/or aPTT ≤ the upper limit of the therapeutic range for intended use.
* Able to provide written informed consent.
* Aged ≥18 years.
* Weight ≥40 kg.
* All male and female Participants who are able to have children must practice effective birth control while on study therapy and for up to 3 months post completion of study therapy. Acceptable forms of birth control for female Participants include: hormonal contraception (implant, injectable contraceptive, transdermal patch, vaginal ring), intrauterine device, tubal ligation or hysterectomy, subject/partner post vasectomy, diaphragm with spermicide, condom with spermicide, or abstinence. Female Participants who become pregnant or suspect pregnancy must immediately notify their doctor. Female Participants who become pregnant will be taken off study. Men who are able to have children must use effective birth control while on the study therapy. Acceptable forms of birth control for male Participants include: vasectomy, condom with spermicide or abstinence. If the male Participant fathers a child or suspects that he has fathered a child while on the study, he must immediately notify his doctor.
* Negative serum or urine beta human chorionic gonadotropin pregnancy test for females of childbearing potential (defined as not postmenopausal for 24 months or no previous surgical sterilization or lactating females) at screening.
* Signed consent to long-term follow-up on protocol PA17-0483 and lab protocols PA17-0577 and LAB02-152.

Exclusion Criteria

* Presence of clinically significant ongoing Grade ≥ 2 toxicity unequivocally associated withthe previous anticancer treatment, as determined by the PI. Toxicities related to priorsurgery, radiation, prior systemic immune checkpoint inhibitors and chemotherapy should be resolved to Grade 1 or below prior to lymphodepletion.
* Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management or not responding to appropriate therapy. Note: Participants with simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
* Known active hepatitis B or C.
* Known human immunodeficiency virus (HIV).
* Presence of active neurological disorder(s).
* Active autoimmune disease within 12 months of enrollment (excluding low-grade psoriasis or well-controlled autoimmune thyroid disease).
* Amyloidosis or POEMS syndrome.
* Symptomatic or uncontrolled central nervous system involvement or signs of cord compression. In the case radiation therapy is indicated, the washout must be at least 14 days.
* Participants must not have any other malignancies within the past 2 years except for in situ carcinoma of any site, adequately treated (without recurrence post resection or post radiotherapy) carcinoma of the cervix or basal or squamous cell carcinomas of the skin, or active non-life-threatening second malignancy that would not, in the investigator's opinion, potentially interfere with the Participant's ability to participate and/or complete this trial. Examples include but are not limited to urothelial cancer Grade Ta or T1 and adenocarcinoma of the prostate treated by active surveillance.
* Presence of any other serious medical condition that may endanger the Participant at investigator's discretion, including but not limited to:
* New York Heart Association Class III or IV heart failure
* Myocardial infarction or stroke ≤ 26 weeks prior to CAR NK cell infusion
* Unstable angina within ≤ 13 weeks prior to CAR NK cell infusion unless the underlying disease has been corrected by procedural intervention (e.g., stent, bypass)
* Severe aortic stenosis
* Uncontrolled arrhythmia. PI approval is required for Participants with arrhythmia who may be included as an exception.
* Congenital long QT syndrome. PI approval is required.
* Documentation, during the screening process, of a QTc > 470 milliseconds by Fredericia criteria (QTcF) based on the average of 3 electrocardiograms (ECGs) taken approximately 1 minute apart and all within 10 minutes of each other. The patient should be reclining for 5 minutes prior to ECGs. Local readings may be used for this exclusion criterion.
* Major surgery < 4 weeks prior to first dose of lymphodepleting chemotherapy.
* Concomitant use of other investigational agents.
* Concomitant use of other anticancer agents.
* Participants receiving systemic steroid therapy at time of enrollment, with an exception for topical, ocular, intranasal, and inhaled corticosteroids, or systemic corticosteroids at an equivalent dose ≤ 10 mg of prednisone daily (physiological substitutive doses are allowed).
* Received antithymocyte globulin within 14 days or alemtuzumab within 28 days of enrollment.
* Participants receiving immunosuppressive therapy.
* Pregnant or breastfeeding.
* Has received a live vaccine within 6 weeks prior to CAR NK cell infusion. Examples of live vaccines include but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza and COVID-19 vaccines for injection are generally killed virusvaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTACAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Johns, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org